CLINICAL TRIAL: NCT04070794
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Study to Investigate Food-effect Bioavailability of Fixed Dose Combination Zemimet® SR Tab. 50/1000 mg (Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg) Under Fed and Fasting Conditions in Healthy Volunteers
Brief Title: Food-effect Bioavailability of Fixed Dose Combination Zemimet® SR Tab. 50/1000 mg Under Fed and Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DMCL008
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — LC15-0444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FDC Zemimet® SR Tab. 50/1000(Fasting) (Active Comparator): Gemigliptin/Metformin Fixed Dose Combination Zemimet® SR Tab. 50/1000 mg (Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg) under fasting condition
  Interventions: Drug: Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg(Fasting)
- FDC Zemimet® SR Tab. 50/1000(Fed) (Active Comparator): Gemigliptin/Metformin Fixed Dose Combination Zemimet® SR Tab. 50/1000 mg (Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg) under fed condition
  Interventions: Drug: Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg(Fed)

INTERVENTIONS:
Drug: Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg(Fasting) — Fasting conditions: Each subject will receive a single dose of fixed dose combination Zemimet® SR Tab. 50/1000 mg with 240±2 mL of 20% glucose solution in drinking water after an overnight fasting for at least 8 hours.
  Arms: FDC Zemimet® SR Tab. 50/1000(Fasting)
Drug: Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg(Fed) — Fed conditions: Each subject will receive a single dose of fixed dose combination Zemimet® SR Tab. 50/1000 mg with 240±2 mL of 20% glucose solution in drinking water at 30 minutes after the start of standardized HFHC breakfast.
  Arms: FDC Zemimet® SR Tab. 50/1000(Fed)

SUMMARY:
A randomized, open-label, single oral dose, one-treatment, two-period, two-sequence, crossover bioavailability study under fed and fasting conditions in healthy Thai volunteers with at least 7 days washout period between the administrations of investigational products of two consecutive periods.

A: Fixed dose combination Zemimet® SR Tab. 50/1000 mg orally administered once without food (fasting conditions) B: Fixed dose combination Zemimet® SR Tab. 50/1000 mg orally administered once with food (fed conditions)

DETAILED DESCRIPTION:
[Objectives] Primary: To investigate the food-effect bioavailability of absorption of gemigliptin/metformin hydrochloride sustained release 50/1000 mg FDC tablet (Zemimet® SR Tab. 50/1000 mg) in healthy subjects under fed and fasting conditions Secondary: To evaluate safety of investigational product under fed and fasting conditions

[Admission and Confinement] Fed conditions: Subjects will be admitted the night before investigational product administration, supervised for at least 8 hours overnight fasting prior to consume standard HFHC breakfast and in-house stay until 24 hours post-dose.

Fasting conditions: Subjects will be admitted a night before investigational product administration, supervised for at least 8 hours overnight fasting prior to dosing and in-house stay until 24 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 to 30.0 kg/m2.
* Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening.
* Non-pregnant woman (negative pregnancy test) and not currently breast feeding.
* Female subjects abstain from either hormonal methods of contraception
* Male subjects who are willing or able to use effective contraceptive
* Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study

Exclusion Criteria:

* History serious hypersensitivity reactions
* History or evidence of clinically significant diseases or any significant ongoing chronic medical illness
* History or evidence of family diabetes
* History or evidence of type 1 diabetes mellitus, diabetic ketoacidosis, diabetic pre-coma
* History or evidence of shock or severe dehydrate or severe infection such as respiratory tract infection, urinary tract infection within 14 days prior to admission in each period
* History or evidence of preceding diarrhea or vomiting within 24 hours prior to admission in each period
* History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse
* History of problems with swallowing tablet or capsule
* Difficulty fasting or consuming standardized meals
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Any condition possibly affecting drug absorption
* Have renal creatinine clearance (Clcr) < 45 mL/min based on serum creatinine results at the screening laboratory test
* 12-lead ECG demonstrating QTc >450 msec, a QRS interval >120 msec or with an abnormality considered clinically significant at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of gemigliptin, LC 15-0636 and metformin | Blood samples (10 mL each) will be collected at time 0.00 (pre-dose; 2x10 mL in duplicate tubes) and at 0.25, 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 24.00 and 48.00 hours post-dose.
  The observed maximum or peak concentration after administration of the drug
AUC0-tlast of gemigliptin, LC 15-0636 and metformin | Blood samples (10 mL each) will be collected at time 0.00 (pre-dose; 2x10 mL in duplicate tubes) and at 0.25, 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 24.00 and 48.00 hours post-dose.
  Area under the concentration-time curve from time zero to the last time where plasma concentration can be measured
AUC0-∞ of gemigliptin, LC 15-0636 and metformin | Blood samples (10 mL each) will be collected at time 0.00 (pre-dose; 2x10 mL in duplicate tubes) and at 0.25, 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 24.00 and 48.00 hours post-dose.
  Area under the concentration-time curve from time zero to infinity by the extrapolation of the rest of AUC from last time where plasma concentration can be measured to time infinity

CONTACTS AND LOCATIONS:
Overall Officials: Uthai Suvanakoot, Principal Investigator — International Bio Service Co., Ltd.

IPD SHARING:
Plan to Share IPD: No